CLINICAL TRIAL: NCT02780713
Title: A Phase I Study to Evaluate the Pharmacokinetic and Safety Profile of AZD9496 Following Single Dose Administration of Different Forms and Formulations in Healthy Subjects
Brief Title: A Study to Assess the Pharmacokinetics and Safety of Different Forms and Formulations of AZD9496 in Healthy Subjects
Acronym: PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6090C00005
Record Dates: First submitted 2016-05-20; First posted 2016-05-23 (Estimated); Results first posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Healthy volunteers; Pharmacokinetics; AZD9496; Safety; Tolerability
MeSH Terms: conditions — Breast Neoplasms | interventions — AZD9496

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD9496 (Experimental): This is a fixed sequence study with 5-sequential treatment periods in healthy volunteers. Each volunteer will receive 5 single doses of AZD9496 in different forms, formulations and doses.
  1. Treatment period 1 will assess AZD9496 Variant A: 100mg.
  2. Treatment period 2 will assess AZD9496 Reference: 100mg.
  3. Treatment period 3 will assess one of AZD9496 Variants, B, C or D: 100mg.
  4. Treatment period 4 will assess one of AZD9496 Variants, B, C or D: 100mg.
  5. Treatment period 5 will assess one of AZD9496 Variants A, B, C or D: *300mg. *Based on a review of PK and safety results from Treatment Periods 1, 3 and 4, a lower dose of 200 mg may be administered in Treatment Period 5
  Interventions: Drug: AZD9496 (Reference); Drug: AZD9496 Variant A; Drug: AZD9496 Variant B; Drug: AZD9496 Variant C; Drug: AZD9496 Variant D

INTERVENTIONS:
Drug: AZD9496 (Reference) — AZD9496 (Reference)
Drug: AZD9496 Variant A — AZD9496 Variant A.
Drug: AZD9496 Variant B — AZD9496 Variant B
Drug: AZD9496 Variant C — AZD9496 Variant C
Drug: AZD9496 Variant D — AZD9496 Variant D

SUMMARY:
This is a phase 1 open label single centre study of AZD9496 administered orally in healthy volunteers. The study design involves single administration of different forms, formulations and doses of AZD9496. The study is designed to investigate these different AZD9496 variants. The study will evaluate the pharmacokinetic profiles and the safety and tolerability of the different forms, formulations and doses of AZD9496

This is a fixed sequence study with 5-sequential treatment periods in healthy volunteers. Each volunteer will receive 5 single doses of AZD9496 in different forms, formulations and doses.

DETAILED DESCRIPTION:
A phase 1, open-label, single centre study to assess the pharmacokinetics, Safety and tolerability of different forms, formulations and doses of AZD9496 in healthy volunteers. This is a fixed sequence study with 5-sequential treatment periods. Each subject will receive 5 single doses of AZD9496 in different forms, formulations and doses.

* Treatment period one will assess AZD9496 Variant A: 100mg.
* Treatment period two will assess AZD9496 Reference form: 100mg.
* Treatment period 3 will assess one of AZD9496 Variants, B, C or D: 100mg.
* Treatment period 4 will assess one of AZD9496 Variants, B, C or D: 100mg.
* Treatment period 5 will assess one of AZD9496 Variants A, B, C or D: *300mg. *Based on a review of pharmacokinetic and safety results from Treatment Periods 1, 3 and 4, a lower dose of 200 mg may be administered in Treatment Period 5.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and/or female subjects aged 18 to 65 years with suitable veins for cannulation or repeated venipuncture.
3. Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating and must be of non-childbearing potential, confirmed at screening by fulfilling 1 of the following criteria: Post-menopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and FSH levels in the post-menopausal range (OR) Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but not tubal ligation
4. Male subjects aged 18 to 39 years must be vasectomized. Male subjects aged 40 to 65 years must either be vasectomized or have no intention of fathering a child for a period of 6 months after receiving the last dose of IMP.
5. Have a body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive, and weigh at least 50 kg and no more than 100 kg, inclusive.
6. Values for AST, ALT, TBL, GGT and ALP must be at or below the upper limit of normal ranges at screening.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
4. Previous history of venous or arterial thromboembolism or thrombophilia.
5. History of endometrial polyps, endometrial cancer, atypical endometrial hyperplasia, or other endometrial disorders unless subjects have undergone total hysterectomy and there is no evidence of active disease (females only).
6. Any clinically significant abnormalities in clinical chemistry (other than Inclusion no.6), hematology, or urinalysis results at screening, as judged by the investigator.
7. Any clinically significant abnormal findings in supine vital signs, after 10 minutes of supine rest, at screening and/or admission to the unit, defined as: (a) Systolic blood pressure < 90 mmHg or ≥ 150 mmHg (b) Diastolic blood pressure < 50 mmHg or ≥ 95 mmHg and (c) Heart rate < 45 or > 90 beats per minute
8. Any clinically important abnormalities in rhythm, conduction or morphology of the resting 12-lead ECG that, as judged by the investigator, that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology or pronounced left ventricular hypertrophy.
9. Prolonged QTcF > 460 ms for females and QTcF > 450 ms for males or family history of long QT syndrome.
10. PR (PQ) interval shortening < 110 ms or evidence of ventricular pre-excitation).
11. PR (PQ) interval prolongation > 240 ms, intermittent second (Wenckebach block while asleep is not exclusive) or third degree AV block.
12. Persistent or intermittent complete bundle branch block with QRS > 120 ms or evidence of pronounced ventricular hypertrophy or pre-excitation.
13. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) antibody.
14. Known or suspected history of drug abuse, as judged by the investigator.
15. Current smokers or those who have smoked or used nicotine products within the 3 months prior to screening.
16. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol, as judged by the investigator.
17. Positive screen for drugs of abuse, alcohol or cotinine at screening or on each admission to the unit.
18. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD9496.
19. Excessive intake of caffeine/xanthine containing drinks or food (e.g., coffee, tea, chocolate), as judged by the investigator.
20. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
21. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life Note: Hormonal replacement therapy is not allowed for females.
22. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening
23. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion is 3 months after the final dose from previous study or 1 month after the last visit of previous study, whichever is the longest. ote: Subjects consented and screened, but not dosed in this study or a previous phase I study, are not excluded.
24. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives
25. Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
26. Subjects who are vegans or have medical dietary restrictions.
27. Subjects who cannot communicate reliably with the investigator.
28. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2016-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ronald Goldwater, Principal Investigator — Parexel
Locations (1):
- Research Site, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the United States (US, 1 site), 14 healthy participants were treated with AZD9496 (1 dose at fasted state) in 5 treatment periods: Formulation Variants A, B & C (doses 1,3, & 4), reference (dose 2) and formulation Variant B (dose 5). Each subject was involved in the study for approximately 10 to 12 weeks.
Pre-assignment Details: A screening period of maximum of -28 days.
Groups:
- Treatment Period 1: Participants received AZD9496 - Variant A (100 mg).
- Treatment Period 2: Participants received AZD9496 - Reference (100 mg).
- Treatment Period 3: Participants received AZD9496 - Variant B (100 mg).
- Treatment Period 4: Participants received AZD9496 - Variant C (100 mg).
- Treatment Period 5: Participants received AZD9496 - Variant B (300 mg).
Period: Period 1: Variant A (100mg)
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Started (Participants received AZD9496 in 5-sequential treatment periods.) | 14 (After washout period participants entered Treatment Period 2.) | 0 (After washout period participants entered Treatment Period 3.) | 0 (After washout period participants entered Treatment Period 4.) | 0 (After washout period participants entered Treatment Period 5.) | 0
Completed (12 participants received and completed treatment and 2 participants withdrew from the study) | 14 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 2: Reference (100mg)
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Started | 0 | 14 | 0 | 0 | 0
Completed (12 participants received and completed treatment and 2 participants withdrew from the study) | 0 | 14 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 3: Variant B (100mg)
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Started | 0 | 0 | 14 | 0 | 0
Completed (12 participants received and completed treatment and 2 participants withdrew from the study) | 0 | 0 | 12 | 0 | 0
Not Completed | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0
Period: Period 4: Variant C (100mg)
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Started | 0 | 0 | 0 | 12 | 0
Completed (12 participants received and completed treatment and 2 participants withdrew from the study) | 0 | 0 | 0 | 12 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 5: Variant B (300mg)
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Started | 0 | 0 | 0 | 0 | 12
Completed (12 participants received and completed treatment and 2 participants withdrew from the study) | 0 | 0 | 0 | 0 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All enrolled participants who received at least one dose of AZD9496.
Arm/Group | All Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.6 (6.22)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 14
  Female | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) for AZD9496 and Its Metabolites at Each Treatment Period.
Description: To evaluate maximum observed plasma concentration (Cmax) for AZD9496 and its metabolites M3 and M5 following administration of different AZD9496 formulations and compare with a reference formulation.
Time Frame: Regular Pharmacokinetic measurement Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 12, hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3), 72 hours post-dose (Day 4) of each treatment period
Population: Safety set with 1 primary PK parameter for AZD9496 calculable for Treatment Period 2 and 1 other period. For AUC 0-inf, a predefined R2adj >0.8 (the goodness of fit parameter for regression estimate of elimination rate constant lambda z used in the AUC 0-inf calculation) was used to determine if the individual AUC estimate was reportable.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Number analyzed (Participants) | 14 | 14 | 12 | 12 | 12
ng/mL
  AZD9496 | 64.85 (73.54) | 381.0 (55.83) | 138.2 (75.35) | 91.83 (52.13) | 550.9 (41.85)
  M3 | 10.30 (98.93) | 62.98 (76.91) | 23.56 (74.30) | 14.47 (39.01) | 98.72 (54.80)
  M5 | 1.102 (85.27) | 7.409 (75.18) | 2.454 (80.35) | 1.520 (42.67) | 11.71 (49.60)

2. Primary Outcome: Pharmacokinetics: Area Under the Curve From Time Zero to Time With Last Observation (AUC0-t) for AZD9496 and Its Metabolites at Each Treatment Period
Description: To evaluate the area under the plasma concentration-curve from time zero to time of last quantifiable concentration (AUC (0-t) of AZD9496 and its metabolites M3 and M5 following administration of different AZD9496 formulations and compare with a reference formulation
Time Frame: Regular Pharmacokinetic measurement: At Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 12, hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3), 72 hours post-dose (Day 4) of each treatment period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Number analyzed (Participants) | 14 | 14 | 12 | 12 | 12
ng*h/mL
  AZD9496 | 383.4 (60.54) | 1207 (53.01) | 677.8 (50.08) | 523.0 (26.77) | 2322 (32.12)
  M3 | 46.71 (124.65) | 196.6 (80.92) | 111.7 (62.00) | 78.23 (65.96) | 411.3 (57.56)
  M5 | 4.872 (98.91) | 23.11 (73.68) | 11.05 (62.20) | 7.614 (57.93) | 46.42 (49.23)

3. Primary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) for Variant A, B and C of AZD9496 Compared to the AZD9496 Reference
Description: To evaluate maximum plasma concentration (Cmax) of capsule variants by comparing with reference AZD9496
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Groups:
- DN Ratio - Variant A (100 mg): Ref (100 mg): Participants received AZD9496 - Variant A (100 mg) in Treatment Period 1.
- DN Ratio - Variant B (100 mg) : Ref (100 mg): Participants received AZD9496 - Variant B (100 mg) in Treatment Period 3.
- DN Ratio - Variant C (100 mg) : Ref (100 mg): Participants received AZD9496 - Variant C (100 mg) in Treatment 4.
Arm/Group | DN Ratio - Variant A (100 mg): Ref (100 mg) | DN Ratio - Variant B (100 mg) : Ref (100 mg) | DN Ratio - Variant C (100 mg) : Ref (100 mg)
Number analyzed (Participants) | 14 | 12 | 12
Ratio | 0.1702 (90.94) | 0.3440 (110.40) | 0.2285 (89.40)
Statistical Analysis 1: Comparison: DN Ratio - Variant A (100 mg): Ref (100 mg); Test type: Superiority; Percentage = 17.02, 95% CI 2-sided [11.79 to 24.58]
Statistical Analysis 2: Comparison: DN Ratio - Variant B (100 mg) : Ref (100 mg); Test type: Superiority; Percentage = 36.28, 95% CI 2-sided [23.84 to 55.20]
Statistical Analysis 3: Comparison: DN Ratio - Variant C (100 mg) : Ref (100 mg); Test type: Superiority; Percentage = 24.10, 95% CI 2-sided [16.84 to 34.48]

4. Primary Outcome: Pharmacokinetics: Area Under the Curve From Time Zero to Time With Last Observation (AUC0-t) for Variant A, B and C of AZD9496 Compared to the AZD9496 Reference
Description: To evaluate area under curve from time zero to time with last observation (AUC0-t) of variants by comparing with reference AZD9496
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Groups:
- AZD9496 - Variant C (100 mg): Participants received this treatment in Treatment Period 4
Arm/Group | DN Ratio - Variant A (100 mg): Ref (100 mg) | DN Ratio - Variant B (100 mg) : Ref (100 mg) | AZD9496 - Variant C (100 mg)
Number analyzed (Participants) | 14 | 12 | 12
Ratio | 0.3175 (46.35) | 0.5227 (50.95) | 0.4033 (33.15)
Statistical Analysis 1: Comparison: DN Ratio - Variant A (100 mg): Ref (100 mg); Test type: Superiority; Percentage = 31.75, 95% CI 2-sided [25.77 to 39.12]
Statistical Analysis 2: Comparison: DN Ratio - Variant B (100 mg) : Ref (100 mg); Test type: Superiority; Percentage = 54.17, 95% CI 2-sided [42.16 to 69.60]
Statistical Analysis 3: Comparison: AZD9496 - Variant C (100 mg); Test type: Superiority; Pecentage = 41.23, 95% CI 2-sided [34.79 to 48.86]

5. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for AZD9496 and Its Metabolites at Each Treatment Period.
Description: To evaluate time to reach maximum observed plasma concentration (Tmax) for AZD9496 and its metabolites M3 and M5 following administration of different AZD9496 formulations and compare with a reference formulation.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 12, hours post-dose on Day 1, 24 and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3), 72 hours post-dose (Day 4) of each treatment period
Population: The PK analysis set consisted of all subjects in the safety analysis set for whom at least 1 of the primary PK parameters for AZD9496 could be calculated for at least Treatment Period 2 and 1 other treatment period, and who had no major protocol deviations thought to impact on the analysis of the PK data.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Number analyzed (Participants) | 14 | 14 | 12 | 12 | 12
Hours
  AZD9496 | 4.25 [1.50 to 5.60] | 2.25 [1.50 to 3.48] | 3.52 [2.50 to 5.03] | 4.25 [2.50 to 5.02] | 4.25 [2.50 to 6.05]
  M3 | 4.50 [2.00 to 5.60] | 2.50 [1.50 to 4.67] | 3.77 [2.98 to 6.02] | 5.00 [3.00 to 5.12] | 4.26 [2.50 to 6.05]
  M5 | 4.50 [2.00 to 5.60] | 2.50 [1.50 to 4.05] | 4.00 [2.50 to 5.50] | 4.99 [3.00 to 5.12] | 4.51 [2.50 to 6.05]

6. Secondary Outcome: Effective Half-life ( t½,Eff) for AZD9496 and Its Metabolites at Each Treatment Period
Description: To evaluate effective half-life (t½,eff), for AZD9496 and its metabolites M3 and M5 following administration of different AZD9496 formulations and compare with a reference formulation.
Time Frame: as for outcome 1
Population: The PK analysis set consisted of all subjects in the safety analysis set for whom at least 1 of the primary PK parameters for AZD9496 could be calculated for at least Treatment Period 2 and 1 other treatment period, and who had no major protocol deviations thought to impact on the analysis of the PK data. Data not available for all participants.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Number analyzed (Participants) | 14 | 14 | 12 | 12 | 12
Hours
  AZD9496: number analyzed (Participants) | 13 | 14 | 10 | 11 | 12
  AZD9496 | 1.34 (0.45) | 1.11 (0.15) | 1.51 (0.68) | 1.56 (0.36) | 1.36 (0.31)
  M3: number analyzed (Participants) | 8 | 14 | 10 | 6 | 10
  M3 | 1.16 (0.36) | 1.09 (0.17) | 2.02 (1.84) | 1.57 (0.47) | 1.28 (0.28)
  M5: number analyzed (Participants) | 9 | 14 | 11 | 9 | 12
  M5 | 1.15 (0.27) | 1.06 (0.15) | 1.54 (0.70) | 1.42 (0.36) | 1.23 (0.26)

7. Secondary Outcome: Metabolite to Parent Ratios (MRAUC0-t, MRCmax, MRAUC) at Each Treatment Period.
Description: To evaluate metabolite to parent ratios (MRAUC0-t, MRCmax, MRAUC) at each treatment period.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Number analyzed (Participants) | 14 | 14 | 12 | 12 | 12
Ratio
  M3 - MRAUC(0-t) | 0.122 (48.12) | 0.163 (30.75) | 0.165 (33.49) | 0.150 (41.38) | 0.177 (30.28)
  M5 - MRAUC(0-t) | 0.013 (33.81) | 0.019 (22.07) | 0.016 (23.06) | 0.015 (32.71) | 0.020 (21.32)
  M3 - MRCmax | 0.159 (37.68) | 0.165 (25.97) | 0.170 (30.68) | 0.158 (36.29) | 0.179 (27.25)
  M5 - MRCmax | 0.017 (30.16) | 0.019 (21.01) | 0.018 (31.23) | 0.017 (33.79) | 0.022 (20.22)
  M3 - MRAUC: number analyzed (Participants) | 0 | 6 | 3 | 0 | 5
  M3 - MRAUC |  | 0.173 (21.11) | 0.172 (7.81) |  | 0.193 (39.07)
  M5 - MRAUC: number analyzed (Participants) | 0 | 9 | 3 | 0 | 5
  M5 - MRAUC |  | 0.020 (14.91) | 0.018 (10.90) |  | 0.021 (26.57)

8. Primary Outcome: Pharmacokinetics: Area Under the Curve From Time Zero to Infinity for Variant A, B and C of AZD9496 Compared to the AZD9496 Reference
Description: To evaluate area under the curve from time zero to time infinity (AUC 0-infinity) of variants by comparing with reference AZD9496
Time Frame: Regular Pharmacokinnetic measurement Pre-dose, 0.5, 1, 1.5, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 12, hours post-dose on Day 1, 24, and 36 hours post-dose (Day 2), 48 hours post-dose (Day 3), 72 hours post-dose (Day 4) of each treatment period
Population: Safety set with 1 primary PK parameter for AZD9496 calculable for Treatment Period 2 and 1 other period. For AUC 0-inf, a predefined R2adj >0.8 (the goodness of fit parameter for regression estimate of elimination rate constant lambda z used in the AUC 0-inf calculation) was used to determine if the individual AUC estimate was reportable. Data not available for all participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Treatment Period 1 | Treatment Period 3 | Treatment Period 4
Number analyzed (Participants) | 1 | 4 | 4
Ratio | NA (NA) — Data for n=1 available. | 0.6186 (37.26) | 0.4055 (48.13)

9. Primary Outcome: Pharmacokinetics: Area Under the Curve From Time Zero to Infinity (AUC 0-infinity) for AZD9496 and Metabolites at Each Treatment Period
Description: To evaluate area under the curve from time zero to infinity (AUC 0-infinity) for AZD9496 and its metabolites
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Number analyzed (Participants) | 14 | 14 | 12 | 12 | 12
ng*h/mL
  AZD9496: number analyzed (Participants) | 1 | 11 | 5 | 5 | 7
  AZD9496 | NA (NA) — Data could not be calculated due to n=1. | 1238 (46.88) | 968.1 (30.12) | 604.7 (18.37) | 2790 (22.97)
  M3: number analyzed (Participants) | 0 | 7 | 7 | 3 | 7
  M3 |  | 253.2 (58.97) | 99.9 (64.10) | 56.9 (30.78) | 420.6 (76.41)
  M5: number analyzed (Participants) | 3 | 12 | 6 | 0 | 6
  M5 | 5.93 (95.53) | 24.09 (76.00) | 11.15 (65.47) |  | 54.84 (47.54)

10. Secondary Outcome: Pharmacokinetics: AUC From Time Zero to 12 and 24 Hours Post-dose for AZD9496 and Its Metabolites at Each Treatment Period
Time Frame: as for outcome 5
Population: Safety set with 1 primary PK parameter for AZD9496 calculable for Treatment Period 2 and 1 other period. For AUC 0-inf, a predefined R2adj >0.8 (the goodness of fit parameter for regression estimate of elimination rate constant lambda z used in the AUC 0-inf calculation) was used to determine if the individual AUC estimate was reportable. Data not available for all participants. Where less than 3 participants contribute data, the PK parameter was not calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Number analyzed (Participants) | 14 | 14 | 12 | 12 | 12
ng*h/mL
  AZD9496 AUC 0-12 Hours | 256.2 (65.67) | 1194 (51.83) | 515.3 (57.4) | 326.3 (36.18) | 1920 (38.5)
  AZD9496 AUC 0-24 Hours: number analyzed (Participants) | 13 | 13 | 11 | 12 | 12
  AZD9496 AUC 0-24 Hours | 299.9 (60.13) | 1306 (44.9) | 614.8 (49.08) | 411.7 (28) | 2130 (36.83)
  M3 AUC 0-12 Hours: number analyzed (Participants) | 8 | 5 | 7 | 7 | 11
  M3 AUC 0-12 Hours | 63.02 (72.17) | 377.3 (23.86) | 91.52 (57.32) | 62.41 (33.9) | 391.6 (46.7)
  M3 AUC 0-24 Hours: number analyzed (Participants) | 5 | 1 | 5 | 6 | 8
  M3 AUC 0-24 Hours | 73.26 (71.57) | NA (NA) — Not calculated as n=1. | 114.9 (47.43) | 91.49 (32.74) | 490.4 (47.82)
  M5 AUC 0-12 Hours: number analyzed (Participants) | 7 | 8 | 6 | 9 | 12
  M5 AUC 0-12 Hours | 6.162 (78.95) | 37.83 (33.76) | 8.646 (74.31) | 5.953 (31.78) | 40.2 (49.71)
  M5 AUC 0-24 Hours: number analyzed (Participants) | 5 | 1 | 5 | 7 | 11
  M5 AUC 0-24 Hours | 7.417 (65.09) | NA (NA) — Not calculated as n=1. | 10.09 (60.5) | 8.32 (27.76) | 46.57 (49.04)

11. Secondary Outcome: Pharmacokinetics: The Terminal Elimination Half-life (t½,λz) for AZD9496 and Its Metabolites at Each Treatment Period
Time Frame: as for outcome 5
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Number analyzed (Participants) | 14 | 14 | 12 | 12 | 12
Hours
  AZD9496: number analyzed (Participants) | 1 | 11 | 5 | 5 | 7
  AZD9496 | NA (NA) — Not calculated as n=1. | 2.59 (1.75) | 8.95 (7.55) | 15.66 (4.47) | 9.65 (3.96)
  M3: number analyzed (Participants) | 2 | 7 | 7 | 3 | 7
  M3 | NA (NA) — Not calculated as n=2. | 1.34 (0.39) | 2.19 (2.13) | 1.89 (0.57) | 3.69 (2.70)
  M5: number analyzed (Participants) | 3 | 12 | 6 | 0 | 5
  M5 | 1.18 (0.47) | 1.89 (1.35) | 1.41 (0.55) |  | 5.06 (2.25)

12. Secondary Outcome: Pharmacokinetics: Apparent Volume of Distribution (Vss/F) of AZD9496 and Its Metabolites at Each Treatment Period
Time Frame: Day 1, Day 2, Day 3 and Day 4
Population: Too few data points available. Data not calculated for Vss/F for M3 and M5 .
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Number analyzed (Participants) | 14 | 14 | 12 | 12 | 12
L
  AZD9496: number analyzed (Participants) | 0 | 11 | 5 | 5 | 7
  AZD9496 |  | 277.5 (127.3) | 1291 (1097) | 3495 (1532) | 920.7 (392.1)
  M3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  M5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Pharmacokinetics: Apparent Oral Clearance (CL/F) of AZD9496 and Its Metabolites at Each Treatment Period
Time Frame: Day 1, Day 2, Day 3 and Day 4
Population: Too few data points available. CL/F not calculated for M3 and M5. Where less than 3 participants contribute data, the PK parameter was not calculated.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Number analyzed (Participants) | 14 | 14 | 12 | 12 | 12
L/h
  AZD9496: number analyzed (Participants) | 1 | 11 | 5 | 5 | 7
  AZD9496 | NA (NA) — Not calculated as n=1. | 80.8 (39.8) | 107.0 (32.7) | 167.5 (30.1) | 110.0 (26.7)
  M3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  M5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Pharmacokinetics: Apparent Terminal Elimination Rate Constant (λz) of AZD9496 and Its Metabolites at Each Treatment Period
Time Frame: Day 1, Day 2, Day 3, Day 4
Population: Too few data points available and so λz not calculated for all participants. Where less than 3 participants contribute data, the PK parameter was not calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: T-1
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Number analyzed (Participants) | 14 | 14 | 12 | 12 | 12
T-1
  AZD9496: number analyzed (Participants) | 1 | 11 | 5 | 5 | 7
  AZD9496 | NA (NA) — Not calculated as n=1. | 0.3132 (58.96) | 0.1236 (183.17) | 0.0459 (31.05) | 0.0777 (46.67)
  M3: number analyzed (Participants) | 2 | 7 | 7 | 3 | 7
  M3 | NA (NA) — Not calculated as n=2. | 0.537 (29.69) | 0.422 (88.14) | 0.380 (34.17) | 0.230 (75.62)
  M5: number analyzed (Participants) | 3 | 12 | 6 | 0 | 6
  M5 | 0.618 (38.36) | 0.426 (55.48) | 0.526 (41.77) |  | 0.154 (65.20)

15. Secondary Outcome: Pharmacokinetics: Mean Residence Time (MRT) of AZD9496 and Its Metabolites at Each Treatment Period
Time Frame: Day 1, Day 2, Day 3, Day 4
Population: Data points not available for all participants. MRT not calculated for M3 and M5 metabolites. Where less than 3 participants contribute data, the PK parameter was not calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5
Number analyzed (Participants) | 14 | 14 | 12 | 12 | 12
Hours
  AZD9496: number analyzed (Participants) | 1 | 11 | 5 | 5 | 7
  AZD9496 | NA (NA) — Not calculated as n=1. | 3.122 (23.77) | 8.992 (107.76) | 19.73 (52.63) | 7.939 (29.73)
  M3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  M5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From enrollment until the final follow-up visit (5 to 7 days after last dose)
Description: Serious adverse events (SAEs) were recorded from the signing of the informed consent and adverse events (AEs) were recorded from enrollment until the final follow-up visit.
  Note: A total of 4 participants reported at least one AE. Of the 4 participants, 1 participant reported two AEs "Rhinorrhoea" and "Body tinea" associated with treatments Variant A and B, respectively.
Arm/Group | Treatment Period 1 | Treatment Period 2 | Treatment Period 3 | Treatment Period 4 | Treatment Period 5 | All Participants
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/12 | 0/12 | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/12 | 0/12 | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 2/14 | 1/14 | 1/12 | 0/12 | 1/12 | 5/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period 1 (N=14) | Treatment Period 2 (N=14) | Treatment Period 3 (N=12) | Treatment Period 4 (N=12) | Treatment Period 5 (N=12) | All Participants (N=14)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Note: Participant who reported "Rhinorrhoea" also reported "Body tinea"
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Note: Participant who reported "Body tinea" also reported "Rhinorrhoea"
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Data from all analysed secondary pharmacokinetic parameters are presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All of the study information and data collected during the study are confidential and the property of AstraZeneca. After completion of the study, the investigator may prepare a joint publication with AstraZeneca. The investigator must undertake not to submit any part of the individual data from this clinical study protocol for publication without prior consent of AstraZeneca at a mutually agreed time.